CLINICAL TRIAL: NCT00850915
Title: Feasibility and Effectiveness of Community Based Isoniazid Preventive Therapy in Kenya
Acronym: IPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KNCV Tuberculosis Foundation (Other)
Collaborators: Stichting Mondiale Tuberculose (SMT) (Unknown); Kenya Medical Research Institute (Other); Division of Leprosy Tuberculosis and Lung Disease, MOPHS, Kenya (Unknown); Centres for Disease Control and Prevention, Kenya. (Other); Ministry of Public Health and Sanitation, Kenya (Other); Kenya National AIDS & STI Control Programme (Other)
Responsible Party: Principal Investigator, Eveline Klinkenberg, senior epidemiologist, KNCV Tuberculosis Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UR-01-2009-IPT-KENYA
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Tuberculosis
Keywords: tuberculosis; community IPT; isoniazid adverse events; tuberculosis incidence
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): in this arm contacts of enrolled TB-HIV index cases were actively approached and screened for TB and offered HIV testing by CHW at their homes
  Interventions: Other: community IPT
- 2 (Other): no interventation was done in this group, they received the regulare care and follow up following NTP guidelines
  Interventions: Other: community IPT

INTERVENTIONS:
Other: community IPT — In the intervention group, the household contacts of enrolled TB/HIV co-infected patient are visited at home by community health workers. Those contacts providing informed consent and considered fit (assessed by simple questionnaire) are assumed not to have active TB and are eligible for IPT. They are offered isoniazid at 300mg (5 mg per Kg for children) once daily for 6 months, regardless of their HIV-status.
  In the control group, in line with routine care, eligible index cases are requested to send their contacts to the clinic for evaluation. Contacts presenting to the clinic will be screened for TB and receive IPT, if under 5 years and when active TB is ruled out as per the current national guidelines.
  All contacts (both intervention and control group) are followed up monthly to assess occurrence of symptoms suggestive of TB.

SUMMARY:
Isoniazid preventive therapy (IPT) is a well studied clinical intervention for primary and secondary prevention of active tuberculosis (TB) after infection with Mycobacterium tuberculosis. It is widely used in industrialized countries in TB outbreak management, focusing on high risk groups such as close contacts in the family, in congregate settings, and in the workplace amongst others. Individuals infected with Human Immunodeficiency Virus (HIV) have a markedly higher risk of acquiring a TB-infection and developing consequently active TB, making HIV-infected individuals a target population for IPT. Studies of IPT in HIV infected persons in the nineties demonstrated the efficacy of IPT in the prevention of active TB in Sub -Saharan Africa and more recent studies suggest that the protective effect remains present in individuals on antiretroviral therapy.

Despite the proven efficacy of IPT this intervention has not been taken up by most HIV and TB control programmes in Africa where the burden of TB/HIV is highest. The reasons for the low uptake of IPT are many and varied but include fears of expansion of isoniazid resistance and subsequently the development of multi -drug resistant TB with widespread use of IPT. Additionally screening protocols for excluding active TB and selecting persons for IPT have not been uniformly agreed upon. There have also been concerns that programmes designed to provide IPT may shift TB control programmes from their primary responsibility of finding and treating active TB. Finally it has been unclear as to which programme, between the HIV and the TB control programme, has the primary responsibility of managing the provision of the IPT intervention.

The World Health Organization and other technical agencies engaged in global TB control have recently re-emphasized the need to scale up IPT. In this proposal we outline an operational research study to evaluate the introduction of IPT at community level and to measure its effectiveness at preventing TB. The study is based on the context of expansion of Community-Based Direct Observed Therapy Short Course (CB-DOTS), home-based care and the concept of HIV prevention with positives (PwPs), where there is a real opportunity to focus on the household as a source of HIV-associated tuberculosis.

The study is designed as a cluster randomized trial. It compares the incidence of TB in household contacts including children under 5 of identified TB/HIV co-infected patients, who received IPT through proactive community intervention and those in a control group where the community was handled in the "usual way". In the intervention group household contacts of index cases of HIV positive, smear positive PTB will be visited at home and consenting contacts will be screened for active TB using a simple questionnaire. Those found to be fit will receive isoniazid 300mg (5 mg per Kg for children) once daily for 6 months, regardless of the HIV-status. Those found not to be fit will be referred for further evaluation at the nearest TB diagnostic centre. In the control group, routine care following national guidelines will be offered. This consists of contact invitation and assessment of eligibility for IPT, especially, in children less than 5 years. Both groups will be followed up monthly through household visits. Follow up will be for a total of 24 months including the six months when IPT is provided.

A confidential HIV screening test will be provided to all consenting contacts in both intervention and control group after appropriate counseling.

The primary outcome is the incidence of TB in the intervention and control household contacts. The difference in incidence between the two groups is a measure of efficacy of the intervention. In addition the efficacy of the intervention will be estimated stratified by HIV status of household contacts if data allows. Secondary outcomes are the incidence of adverse events, the incidence of TB-related symptoms, measures on the uptake of IPT (proportion of contacts starting and discontinuing IPT, treatment adherence) and programmatic indicators, i.e. percentage of persons eligible for IPT and resources needed.

ELIGIBILITY:
Index cases

* New sputum smear positive pulmonary tuberculosis (PTB) patients initiating treatment for TB
* HIV infected
* Resident in the catchment area of the TB diagnostic facility
* Written informed consent
* Age equal or greater than 15 years.

Contacts

* Household contacts of a HIV infected smear positive PTB
* No plans to relocate to another area for at least the next two years
* Asymptomatic (Fit) with no cough in last 2 weeks, fever, weight loss (or failure to gain weight in children), haemoptysis or chronic diarrhea at least for the last one month.
* Written informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1259 (Actual)
Dates: Start 2009-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
incidence of TB in household contacts | 12, 18, 24 months

SECONDARY OUTCOMES:
incidence of adverse events in household contacts | 12, 18, 24 months
incidence of TB-related symptoms in household contacts | 12, 18, 24 months
proportion of household contacts starting IPT | 12, 18, 24 months
proportion of household contacts discontinuing IPT | 12, 18, 24 months
proportion of household contacts adhering to IPT treatment | 12, 18, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Chakaya, MD, Principal Investigator — Centre for Respiratory Diseases Research, Kenya Medical Research Institute; Eveline Klinkenberg, PhD, Principal Investigator — KNCV Tuberculosis Foundation, the Netherlands
Locations (18):
- Kenya (18):
  - Makuyu H/C, Makuyu-Muranga, Central
  - Huruma Lions -Central district, Nairobi, Nairobi North
  - Kangemi HC, Nairobi, Nairobi North
  - Blue House, Mathare, Nairobi, Nairobi South
  - Jericho HC, Nairobi, Nairobi South
  - Kibera AMREF, Nairobi, Nairobi South
  - MMM, Mukuru, Embakasi, Nairobi, Nairobi South
  - Pumwani Majengo H/C, Nairobi, Nairobi South
  - Remand H/C, Nairobi, Nairobi South
  - Soweto Kayole, Embakasi, Nairobi, Nairobi South
  - KAPSABET District Hospital, Kapsabet-Nandi, North Rift
  - NYALENDA, Kisumu District, Nyanza North
  - Kadem leprosy, Migori, Migori District, Nyanza South
  - Muhuru Health centre, Migori, Migori District, Nyanza South
  - Awendo SDH, Rongo District, Nyanza South
  - Lanet, Nakuru, RVS
  - Nakuru West, Nakuru, RVS
  - Narok District Hosp, Narok, RVS